CLINICAL TRIAL: NCT00621790
Title: Efficacy of Fenoldopam in Reducing the Need for Renal Replacement Therapy After Cardiac Surgery. A Randomized Controlled Study.
Brief Title: Fenoldopam and Acute Renal Failure
Acronym: FENO HSR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Head of Research, Anesthesia and Intensive Care Department, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GO/URC/ER/mm 64/DG
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Acute Renal Failure
Keywords: fenoldopam; acute renal failure; renal replacement therapy; mortality; cardiac surgery; cardiac anesthesia; intensive care unit
MeSH Terms: conditions — Acute Kidney Injury | interventions — Fenoldopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fenoldopam (Experimental): Fenoldopam 0.1 ug/kg/min (from 0.025 to 0.3 ug/kg/min) for up to 4 days
  Interventions: Drug: fenoldopam
- Placebo (Placebo Comparator): Placebo (normosaline), continuous perfusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fenoldopam — fenoldopam 0.1 ug/kg/min (from 0.025 to 0.3 ug/kg/min)for up to 4 days
  Other Names: corlopam
  Arms: Fenoldopam
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Patients undergoing cardiac surgery could develop postoperative acute renal failure requiring renal replacement therapy.

Fenoldopam, already used for patients with hypertensive emergencies, could improve renal function in critically ill patients with or at risk for acute renal failure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* who underwent cardiac surgery
* have Risk of Acute Renal Failure (R of RIFLE score)

Exclusion Criteria:

* glaucoma
* already on renal replacement therapy
* study drug in the past 30 days
* inclusion in other protocols

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2008-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of patients requiring Renal Replacement Therapy | participants will be followed for the duration of intensive care unit stay, an expected average of one week

SECONDARY OUTCOMES:
Number of dead patients. | Participants will be followed for 1 year.

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - A.O. Universitario Policlinico S.Orsola Malpighi, Bologna
  - Pres.Ospedal. Spedali Civili Brescia - Brescia, Brescia
  - Azienda Ospedaliera Universitaria "Mater Domini" Catanzaro, Catanzaro
  - Azienda Ospedaliero Universitaria Careggi - Firenze, Florence
  - Città di Lecce Hospital GVM Care and Research Lecce, Lecce
  - Villa Maria Cecilia di Cotignola, Lugo Di Ravenna
  - Azienda Ospedaliera Papardo - Messina, Messina
  - Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia, Milan
  - Azienda Ospedaliera Vincenzo Monaldi - Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera di Perugia - Policlinico Monteluce(Osp. S.Maria della Misericordia), Perugia
  - Azienda Ospedaliero Universitaria Pisana - Pisa, Pisa
  - A.O.Universitario Policlinico Tor Vergata - Roma, Roma
  - Ospedale Civile SS Annunziata di Sassari, Sassari
  - Azienda Ospedaliera Universitaria Senese (Policlinico S.Maria alle Scotte), Siena
  - Azienda Ospedaliera San Giovanni Battista Molinette di Torino, Torino
  - Ospedale Mauriziano Umberto I di Torino, Torino
  - Ospedale S.Maria di Ca' Foncello, Treviso
  - Azienda Ospedaliera Universitaria Santa Maria della Misericordia, Udine

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014
- [Derived] Bove T, Zangrillo A, Guarracino F, Alvaro G, Persi B, Maglioni E, Galdieri N, Comis M, Caramelli F, Pasero DC, Pala G, Renzini M, Conte M, Paternoster G, Martinez B, Pinelli F, Frontini M, Zucchetti MC, Pappalardo F, Amantea B, Camata A, Pisano A, Verdecchia C, Dal Checco E, Cariello C, Faita L, Baldassarri R, Scandroglio AM, Saleh O, Lembo R, Calabro MG, Bellomo R, Landoni G. Effect of fenoldopam on use of renal replacement therapy among patients with acute kidney injury after cardiac surgery: a randomized clinical trial. JAMA. 2014 Dec 3;312(21):2244-53. doi: 10.1001/jama.2014.13573. PMID 25265449